CLINICAL TRIAL: NCT02899559
Title: Messages and Plans to Increase Gym Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 825574
Record Dates: First submitted 2016-08-31; First posted 2016-09-14 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Participants will fill out a brief Qualtrics survey which will expose them to one of three message conditions. The control group will read only summary information about the David Pottruck Health and Fitness Center.
  Interventions: Behavioral: Message
- Nudge Message (Experimental): Participants will fill out a brief Qualtrics survey which will expose them to one of three message conditions. The nudge message encourages participants to make a plan for when they will exercise at the gym during the next week.
  Interventions: Behavioral: Message
- Boost Message (Experimental): Participants will fill out a brief Qualtrics survey which will expose them to one of three message conditions. Those in the Boost condition will also have summary information about the Pottruck gym but will also be given information about why an implantation intention is an effective way to attain long term goals. They will also be given a prompt to form an implementation intention.
  Interventions: Behavioral: Message

INTERVENTIONS:
Behavioral: Message — Participants will receive one of three messages at the end of a survey, two of which are experimental messages and one of which is a control message.

SUMMARY:
This primary object of this study is to test to the hypothesis that the both the nudge and boost messages will increase short term gym utilization relative to the control condition but that only the boost message will increase long-term gym utilization.

Non-technical summary: College students will receive one of three messages about exercise. Their card swipe data as a measure of gym utilization will be tracked as an assessment of the effect of those messages.

DETAILED DESCRIPTION:
Our study uses a survey methodology. Within the survey, participants are randomly assigned to experimental conditions. After completion of the survey, participants' real-world behavior is assessed via gym card swipe data.

Within the survey, an experimental quantitative three group design will be used to answer our research question. Thus, our independent variable has three levels: the control message, the nudge message, and the boost message. Our dependent variable will be collected gym card swipes over the semester.

The three experimental message conditions will be delivered within the questionnaire that participants complete. The control group will read only summary information about the David Pottruck Health and Fitness Center. Participants in the nudge condition will read a similar summary but will also be given a prompt to form an implementation intention. Those in the Boost condition will also have summary information about the Pottruck gym but will also be given information about why an implantation intention is an effective way to attain long term goals. They will also be given a prompt to form an implementation intention.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergraduates at the University of Pennsylvania

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Gym Utilization Over the Course of a Semester | Up to 4 months
  We will collect gym card swipes over the course of a single-academic semester at the University of Pennsylvania.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Milkman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States